CLINICAL TRIAL: NCT06607978
Title: Relationship of Noninvasive Assessment of Central Blood Pressure With 10 Years Atherosclerotic Cardiovascular Disease in Subclinical Hypothyroidism
Brief Title: Relationship of Noninvasive Assessment of Central BP With 10 Years Atherosclerotic CVD in Subclinical Hypothyroidism
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Abdelhameed Saber, Principal investigator, Assiut University
Other Study IDs: Central BP and hypothyroidism
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Subclinical hypothyroïdism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with subclinical hypothyroidism admitted to internal medicine department.: patients with subclinical hypothyroidism admitted to internal medicine department.
- healthy match individual .: healthy match individual

SUMMARY:
verify Relationship of noninvasive assessment of central arterial blood pressure with 10 years Atherosclerotic Cardiovascular disease (ASCVD) in Subclinical hypothyroidism

DETAILED DESCRIPTION:
Subclinical hypothyroidism (SCH), characterized by elevated thyrotropin (TSH) levels with normal free thyroxine (T3,T4) concentrations, is a prevalent disorder affecting approximately 10% of the adult population. It has been increasingly recognized for its potential impact on cardiovascular health. A 10-year follow-up study highlighted a significant association between elevated serum TSH levels and increased cardiovascular (CV) risk, independent of conventional risk factors. And it demonstrated its association with hypercholesterolemia and atherosclerosis as the leading risk of CVD. Moreover, in a recent meta-analysis, subclinical hypothyroidism was shown actually be correlated with an increased risk of CVD and mortality.

Monitoring thyroid function underscores the potential importance of cardiovascular (CV) risk assessment, for patients with subclinical hypothyroidism (SCH). Incorporating thyroid function tests, such as TSH and free thyroxine (FT4) levels, alongside non-invasive central arterial blood pressure monitoring, provides a comprehensive understanding of a patient's CV risk. This integrated approach enables early identification and targeted interventions, ultimately improving patient outcomes and reducing the incidence of CVD among those with SCH.

One of the earliest functional changes underlying ASCVD is Arterial stiffening it reflects a variety of pathologies, including atherosclerosis. As an important determinant of cardiovascular health, arterial stiffness can contribute to increased blood pressure and reduces vessels' capacity to buffer the pulsatile flow when the heart contracts, which are significant risk factors for predicting ASCVD.

For continuous non-invasive central arterial blood pressure monitoring, the auscultatory method or The Oscillometric technique can be used. These methods provide valuable insights into the health of the central arteries, which are crucial in understanding the cardiovascular risk profile of patients with SCH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Both sex

Exclusion Criteria:

* Patients had thyroidectomy operation
* Patients with a history of encompassing acute coronary syndrome (ACS).
* Myocardial infarction (MI).
* Coronary heart disease (CHD).
* Cerebrovascular diseases or other arterial revascularization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Full Personal history will include:
  Demographic data age, sex, material status, smoking history, residence (rural, urban) ,presence of previous medical disease (DM ,HTN, cardiac ,renal disease).
  Full medical history will include Duration of the disease, history of treatment intake ,history of autoimmune disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assess the extent to which subclinical hypothyroidism is associated with atherosclerotic cardiovascular disease | 2025
  the extent to which subclinical hypothyroidism is associated with atherosclerotic cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal, Doctor, Study Director — Dr/ Mohamed Faisal El Adway